CLINICAL TRIAL: NCT02017392
Title: A Randomized Controlled Study of Compound Lidocaine Cream to Prevent Postoperative Agitation in Patients With Endotracheal Intubation for General Anesthesia
Brief Title: A RCT of Compound Lidocaine Cream to Prevent Postoperative Agitation in Patients With Endotracheal Intubation for GA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yanni Wang, student, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: [2013]2-85
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Postoperative Agitation of Patients
Keywords: postoperative agitation; endotracheal intubation; general anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Compound Lidocaine Cream (Experimental): The cuff of endotracheal tube is covered by 1-2g compound lidocaine cream before the general anesthesia.
  Interventions: Drug: Compound Lidocaine Cream
- blank control (No Intervention): No intervention.

INTERVENTIONS:
Drug: Compound Lidocaine Cream — Compound Lidocaine Cream ,1-2 grams per person.
  Arms: Compound Lidocaine Cream

SUMMARY:
The purpose of this study is to determine whether the compound lidocaine cream is effective in preventing postoperative agitation in patients with endotracheal intubation for general anesthesia.

DETAILED DESCRIPTION:
This is a randomized controlled study. Some parameters were provided by preliminary test, provided theα=0.05,and β=0.20, the sample size can be estimated to be 2000 by the Open Epi Version 2.Patients will be recruited on the basis of predefined criterias. A researcher will take charge of the recruitment. Participants provide written consent and no financial incentives are provided. They are divided into experimental group and control group randomly. We need to collect their basic information including ages, genders, heights, weights, underlying diseases, surgical procedures and levels classified by ASA. Blood pressure, heart rate and other vital signs during the tube drawing process will be recorded. All the contents needed to be recorded had been compiled into a watch list with detailed instructions for filling in. All the personal information and observation records of participants will be kept in secret and only used for research. Developing standard operating procedure and training all the researchers. A third party will assess the accuracy, completeness and representativeness of registry data. Experimental data will be analysed with the help of statisticians.

ELIGIBILITY:
Inclusion Criteria:

* aged over 18
* selective operation patients with endotracheal intubation for general anesthesia

Exclusion Criteria:

* highly sensitive to local anesthetics of amide derivatives or anything else in compound lidocaine cream
* congenital or idiopathic methemoglobinemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2013-12; Primary Completion 2014-03 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Vital signs like blood pressure and heart rates during extubation. | an hour

SECONDARY OUTCOMES:
The cough reflex and breath holding during extubation. | an hour

OTHER OUTCOMES:
Application of antihypertensive drugs | an hour

CONTACTS AND LOCATIONS:
Overall Officials: Xun Liu, Associate Professor, Study Chair — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The third affiliated hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Batai I, Bogar L, Juhasz V, Batai R, Kerenyi M. A comparison of the antimicrobial property of lidocaine/prilocaine cream (EMLA) and an alcohol-based disinfectant on intact human skin flora. Anesth Analg. 2009 Feb;108(2):666-8. doi: 10.1213/ane.0b013e31818f887e. PMID 19151306
- [Background] Sawyer J, Febbraro S, Masud S, Ashburn MA, Campbell JC. Heated lidocaine/tetracaine patch (Synera, Rapydan) compared with lidocaine/prilocaine cream (EMLA) for topical anaesthesia before vascular access. Br J Anaesth. 2009 Feb;102(2):210-5. doi: 10.1093/bja/aen364. PMID 19151049
- [Derived] Lv L, Yan L, Liu X, Chen M. Effectiveness of lidocaine/prilocaine cream on cardiovascular reactions from endotracheal intubation and cough events during recovery period of older patients under general anesthesia: prospective, randomized placebo-controlled study. BMC Geriatr. 2020 May 4;20(1):157. doi: 10.1186/s12877-020-01567-y. PMID 32366224